CLINICAL TRIAL: NCT06607016
Title: An Open-Label, Single-Arm Phase II Clinical Trial to Evaluate the Initial Efficacy, Safety, Pharmacokinetics, Pharmacodynamics and Immunogenicity of KJ103 for the Treatment of Patients With Anti-Glomerular Basement Membrane Disease
Brief Title: A Clinical Trial With KJ103 in Anti-GBM Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Bao Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHBJ-KJ103-002
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Anti-Glomerular Basement Membrane Disease
MeSH Terms: conditions — Anti-Glomerular Basement Membrane Disease | interventions — Injections; Cyclophosphamide; Glucocorticoids; Plasma Exchange

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): KJ103 +SOC(SoC consists of a standardized combination of PE, Cyclophosphamide, and glucocorticoids)
  Interventions: Drug: KJ103 for Injection; Drug: Cyclophosphamide; Drug: Glucocorticoids; Procedure: Plasma exchange (PE)

INTERVENTIONS:
Drug: KJ103 for Injection — Subjects will administered KJ103 intravenously on D1 and adjunctively on D8
Drug: Cyclophosphamide — Hence treatment prevents formation of new anti-GBM antibodies.
Drug: Glucocorticoids — Glucocorticoids inhibit the inflammation process.
Procedure: Plasma exchange (PE) — PLEX removes the patient's pathogenic anti-GBM antibodies, by replacement of deficient plasma with a replacement fluid.

SUMMARY:
An open-label, single-arm Phase II study to evaluate the preliminary efficacy, safety, pharmacokinetics, pharmacodynamics and immunogenicity of KJ103 in patients with anti-GBM disease.

DETAILED DESCRIPTION:
Anti-glomerular basement membrane (GBM) disease is a severe, rare autoimmune disorder with an internationally reported incidence of 0.5-1/1 million. It is defined as a vasculitis in which anti-GBM antibodies affect glomerular capillaries, pulmonary capillaries or both. Pulmonary involvement leads to pulmonary haemorrhage and renal involvement can lead to glomerulonephritis with necrosis and crescents.

Anti-GBM disease is a severe autoimmune disorder characterised by rapidly progressive glomerulonephritis and positive anti-GBM antibodies. Antibodies can be found in the circulation and deposited in the lungs and kidneys, mediating renal injury through complement activation and recruitment of inflammatory cells. If left untreated, the vast majority of patients will progress to end-stage renal disease (ESRD) or die from pulmonary haemorrhage. Early detection and measures to reduce anti-GBM antibody levels have the potential to alter prognosis and protect renal function. Unfortunately, many patients with anti-GBM disease are diagnosed late and renal function is not restored even with an aggressive treatment regimen of plasma exchange (PE) combined with immunosuppression. Current KDIGO (Kidney Disease Improving Global Prognosis Organisation) guidelines state that the clinical treatment of anti-GBM disease is a combination of glucocorticoids, cyclophosphamide and PE. Despite treatment, patients continue to produce anti-GBM antibodies in their bodies. Rebound anti-GBM antibodies are usually indicative of adverse renal outcomes and PE must be initiated to remove the rebound antibodies.PE is an effective means of removing circulating anti-GBM antibodies, but only removes about 1/3 of the percentage per treatment, so multiple treatments are required to achieve complete removal.

This is a single-arm Phase II study designed to evaluate the preliminary efficacy, safety, pharmacokinetics, pharmacodynamics and immunogenicity of KJ103 in patients with anti-GBM disease. The trial is expected to enrol 9 to 12 subjects who will receive KJ103 treatment.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged ≥18 years, both sexes.
2. Diagnosed with anti-GBM disease. Positive anti-GBM antibodies at screening, with or without ANCA antibody positivity.
3. With or without symptoms of haematuria and proteinuria.
4. Patients of childbearing potential who do not plan to have children during the study and for 6 months after the end of the study, or who are using effective contraception during sexual intercourse.

Exclusion criteria:

1. Anuria for more than 24 hours prior to the first dose.
2. Diagnosis of anti-GBM disease more than 14 days prior to first dose.
3. Moderate to severe pulmonary haemorrhage requiring mechanical ventilation during the screening period, including those occurring within two weeks prior to signing the informed consent form.
4. Severe renal disease not caused by anti-GBM disease, such as lupus nephritis, which, in the opinion of the investigator, makes them unsuitable for participation in this study.
5. Pregnant or breastfeeding at the time of screening.
6. Have a serious underlying medical condition other than anti-GBM disease, such as infection, autoimmune disease, respiratory disease, cardiovascular disease, central nervous system disease, etc., that the investigator deems unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Renal function | day 90, day 180
  Proportion of subjects with renal function after KJ103 administration.

SECONDARY OUTCOMES:
Adverse events | day 180
  Assessing the incidence and severity of adverse events (AEs) and serious adverse events (SAEs) via the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Proportion and number of subjects requiring PE | day 180
  Proportion and number of subjects requiring PE after KJ103 administration.
Anti-GBM antibodies | day 180
  Number of days positive for anti-GBM antibodies after KJ103 administration.
Immunogenicity | day 180
  Immunogenicity of KJ103 (Anti-KJ103 antibody) in patients with anti-GBM disease.
eGFR and change from baseline. | Day28, Day60, Day90, Day120, Day150, Day180
  Estimated glomerular filtration rate (eGFR). Glomerular filtration rate is an estimate of the amount of ultrafiltrate produced by each side of the kidney per unit of time and is an indicator of kidney function.
Pharmacokinetics of KJ103 (Cmax) | day 7
  Maximum observed serum concentration of KJ103 following dosing (Cmax)
Pharmacokinetics of KJ103 (AUC) | day 7
  Area under the serum concentration versustime curve (AUC)
Pharmacokinetics of KJ103 (t1/2) | day 7
  Half-life of KJ103
Pharmacokinetics of KJ103 (CL) | day 7
  Clearance(CL) is a measure of the ability of the body to clear KJ103
Pharmacokinetics of KJ103 (Vz) | day 7
  Vz = Volume of distribution during the elimination phase
Pharmacodynamic profile (Serum IgG levels) | day 180
  Serum IgG levels after KJ103 dosing
Pharmacodynamics-Anti neutrophil cytoplasmic antibodies (ANCA) | day 180
  Serum Anti neutrophil cytoplasmic antibodies (ANCA) levels after KJ103 dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China